CLINICAL TRIAL: NCT03649048
Title: Randomized Trial Comparing Low-Dose Weekly to High-Dose Cisplatin Concurrent With Radiation for Locally Advanced Head and Neck Cancer.
Brief Title: Low-Dose Weekly vs High-Dose Cisplatin
Acronym: RADIO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Cisplatin HD vs LD
Record Dates: First submitted 2018-06-29; First posted 2018-08-28 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Locally Advanced Head and Neck Squamous Cell Carcinoma
MeSH Terms: interventions — Cisplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARM 1: High-Dose Cisplatin days 1, 22 & 43 with radiotherapy (Active Comparator)
  Interventions: Drug: High-Dose Cisplatin; Radiation: Radiotherapy
- ARM 2: Low-Dose Cisplatin Q 1 wk + radiotherapy (Active Comparator)
  Interventions: Drug: Low-Dose Cisplatin; Radiation: Radiotherapy

INTERVENTIONS:
Drug: High-Dose Cisplatin — Intravenous administration of High-Dose Cisplatin
  Arms: ARM 1: High-Dose Cisplatin days 1, 22 & 43 with radiotherapy
Drug: Low-Dose Cisplatin — Intravenous administration of Low-Dose Cisplatin
  Arms: ARM 2: Low-Dose Cisplatin Q 1 wk + radiotherapy
Radiation: Radiotherapy — Participating centres are to follow their local radiation treatment planning and delivery techniques.

SUMMARY:
This study is a prospective open-label randomized clinical trial. Following informed consent eligible LASCCHN patients (n=100) planned for CRT will be stratified by tumor p16 status and then randomized in a 1:1 fashion to either concurrent HD cisplatin or concurrent weekly LD cisplatin.

DETAILED DESCRIPTION:
Human papilloma virus-related oropharynx cancer is increasing in incidence and is now the most common indication for LASCCHN CRT. It more commonly affects younger patients without other comorbidities and is associated with high rates of cure. This creates a survivorship dilemma, as these patients suffer a greater and more prolonged impact from chronic treatment effects such as hearing loss on their HRQOL. Furthermore, this cohort of patients is more likely to be engaged in contributing to societal and economic productivity for a more prolonged period of time. Minimizing long term side effects through strategies to better individualize treatment has been recognized as a priority by the US NIH.

Efforts to identify risk factors for cisplatin toxicity have been previously reported in pediatric cancer patients. Pussegoda and colleagues identified greater risk of hearing loss with cisplatin in children who carried single nucleotide polymorphisms (SNPs) in thiopurine S-methyltransferase (TPMT) and catechol-O-methyltransferase (COMT) genes. However, the role of these genes in predicting ototoxicity risk has remained controversial with both confirmatory and conflicting reports. Two independent studies identified SNPs in the gene acylphosphatase 2 (ACYP2) as being predictive of ototoxicity in pediatric populations. Additional studies have implicated drug transporters involved in cisplatin disposition including the multidrug and toxin extrusion protein 1 (MATE1) to be associated with platinum response and toxicities. In vitro experiments and know-out studies identified cisplatin as a substrate of MATE1. To date, there remains a paucity of data investigating the association between genetic factors and hearing loss in adult LASCCHN patients. A prospective cohort study conducted at LHSC in collaboration with Dr. Richard Kim studied 206 adult LASCCHN patients receiving CRT with cisplatin and identified four independent risk factors for cisplatin-related hearing loss. Risk of hearing loss was increased with the presence of COMT SNPs (HR = 1.75; 95% CI, 1.17 - 2.52) while MATE1 reduced the risk (HR = 0.46; 95% CI, 0.26 - 0.84). The risk of hearing loss was reduced with cisplatin administered on a weekly low dose (LD) compared to a HD schedule. PFS and OS were similar between SNP cohorts and patients treated with weekly LD cisplatin and HD cisplatin regimens. To validate these results and confirm benefits on the pragmatic endpoint of hearing-related QOL, the investigators propose a prospective randomized clinical trial comparing HD and weekly LD cisplatin.

Opinion leaders such as the National Comprehensive Cancer Network guidelines endorse the use of weekly LD cisplatin as a reasonable alternative to HD cisplatin when administered concurrently with radiation. While the study conducted at LHSC observed weekly LD patients had reduced ototoxicity with similar efficacy compared to HD patients, there is no randomized control trial data in LASCCHN to support this practice. Current American Society of Clinical Oncology (ASCO) guidelines support HD cisplatin in this setting based strength of evidence. Therefore, the optimal schedule and dosing of cisplatin when administered as part of CRT in the curative intent treatment of patients with LASCCHN remains unresolved supporting clinical equipoise as to which constitutes the "best" approach.

The investigators primary hypothesis is that LD weekly cisplatin 40 mg/m² is associated with reduced frequency of severe hearing loss and improved hearing-related QOL when compared to conventional HD cisplatin 100 mg/m² days 1, 22 & 43 (control arm) in LASCCHN patients treated with CRT. Furthermore, the investigators hypothesize that a significant proportion of the risk of cisplatin-related hearing loss is attributable to individual differences in pharmacogenomics factors affecting cisplatin disposition that could be identified prior to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Willing and able to provide written informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Histologically or cytologically confirmed squamous cell carcinoma
* Primary tumor site includes oral cavity, oropharynx, nasal cavity, salivary glands (excluding parotid), hypopharynx, or larynx and primary unknown
* Patients must be deemed suitable for HD cisplatin therapy based on tumor characteristics, clinical condition and comorbidities in the judgement of the treating medical oncologist.
* Patients must be planned to receive radical intent radiation treatment based on clinical condition, comorbidities and tumor characteristics in the judgment of the treating radiation oncologist
* Adequate organ and marrow function independent of transfusion for at least 7 days prior to randomization defined as:

  * Hemoglobin > 80 g/L; Absolute neutrophil count >1.5x10⁹ /L, platelets >100x10⁹/L; Bilirubin < 35 umol/L; AST or ALT < 3 x the upper limit of normal; Calculated creatinine clearance (as determined by Cockcroft- Gault) > 50 ml/min

Males:

Creatinine Clearance = Weight (kg) x (140 - Age) (mL/min) 72 x serum creatinine (mg/dL)

Females:

Creatinine Clearance = Weight (kg) x (140 - Age) x 0.85 (mL/min) 72 x serum creatinine (mg/dL)

* Patient must be assessed at head and neck cancer multidisciplinary clinic (with assessment by radiation oncologist and surgeon) and presented at multidisciplinary tumor board prior to randomization.

Exclusion Criteria:

* Serious medical comorbidities or other contraindications to radiotherapy and/or chemotherapy.
* Prior history of head and neck cancer within 5 years.
* Nasopharyngeal primary confirmed or suspected.
* Severe hearing loss as determined clinically Pre-existing use of hearing aids.
* Peripheral neuropathy .grade 2 (CTCAE v4.02).
* Prior or planned neoadjuvant chemotherapy prior to CRT.
* Prior head and neck radiation at any time.
* Distant metastatic disease.
* Inability to attend full course of radiotherapy or follow-up visits.
* Prior invasive malignant disease unless disease-free for at least 5 years or more, with the exception of non-melanoma skin cancer or in-situ carcinoma.
* Unable or unwilling to complete QOL questionnaires.
* Pregnant or lactating women.
* Unable to use dual method of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-11-05 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Hearing related quality of life (QOL) | 1-year post start of treatment
  Assessed with the Hearing Handicap Inventory for Adults (HHIA) Questionnaires. Scored by a points system. The higher the points the more significant the hearing handicap.
Hearing related quality of life (QOL) | 1-year post start of treatment
  Assessed with the Hearing Handicap Inventory for the Elderly (HHIE). Scored by a points system. The higher the points the more significant the hearing handicap.
Compare Incidence of > Grade 2 hearing loss | At 1 year post start of treatment
  A comprehensive audiological examination including case history, otoscopy, behavioural and physiological auditory measures will be conducted prior to an ototoxic drug administration. Subsequent audiology testing will be performed at 3, 6 and 12 months post-start of treatment.
Compare Incidence of > Grade 1 hearing loss | At 1 year post start of treatment
  Will be scored according to the CTCAE v4.02 (Common Terminology Criteria for Adverse Events)

SECONDARY OUTCOMES:
Proportion of patients recommended for hearing amplification | at year 1 post start of treatment
  This information will be specified on the audiology report and collected on the CRF
Compare incidence of > grade 2 hearing loss | At 6 months and at 1 year post start of treatment
  This information will be specified on the audiology report and collected on the CRF
Change in Health related Quality of Life (HRQOL) | At 1 year post start of treatment
  Measured using the EORTC (European Organisation for Research and Treatment of Cancer) QLQ H&N35 (Quality of Life Questionnaire Head & Neck). According to the EORTC scoring guidelines All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Incidence of > Grade 3 treatment-related neuropathy | At baseline, day 21 and day 42
  Measured using the CTCAE Version 4.02 (Common Terminology Criteria for Adverse Events)
Change in neuropathy-associated QOL | At year 1 post start of treatment
  FACT/GOG-Ntx-4 questionnaire subscale (Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity version 4 subscale). According to the FACT-GOG scoring guidelines Higher scores for the scales and subscales indicate better quality of life.
Incidence of any treatment related nephropathy | A baseline, day 21 and day 42
  Measured using the CTCAE Version 4.02
Prevalence of persistent > Grade 3 nephropathy | At 1 year post start of treatment
  Measured using the CTCAE Version 4.02
Evaluate the validity of MATE1 SNPs as a predictor of ototoxicity | At baseline
  Mutational status will be analyzed on samples collected at baseline
Evaluate the validity of COMT SNPs as a predictor of ototoxicity | At baseline
  Mutational status will be analyzed at baseline
Change in Health related Quality of Life (HRQOL) | At 1 year post start of treatment
  Measured using the EORTC (European Organisation for Research and Treatment of Cancer) QLQ-30 (Quality of Life Questionnaire). According to the EORTC scoring guidelines All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.

OTHER OUTCOMES:
Overall Survival | Captured annually starting at a year post start of treatment and continued for up to 5 years following date of randomization.
  Defined as time from randomization to death from any cause
Progression-free Survival | Captured annually starting at a year post start of treatment and continued for up to 5 years following date of randomization.
  Defined as time from randomization to disease progression at any site or death.
Locoregional control | Captured annually starting at a year post start of treatment and continued for up to 5 years following start of treatment.
  Defined as local if within the zone of the primary tumour, and as regional if occurring elsewhere including neck lymph nodes.
Cost-effectiveness analysis | At 1 year post start of treatment
  Using the EQ-5D-5L questionnaire(EuroQol 5 level questionnaire). The EQ-5D-5L descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. Patient is asked to indicate their health by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Radiation doses to the cochlea | At 1 year post-start of treatment.
  To analyze the relationship between cochlear dose and hearing endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Kuruvilla, MD, Principal Investigator — London Health Sciences Centre, London Regional Cancer Program
Locations (3):
- Canada (3):
  - Juravinski Cancer Centre, Hamilton, Ontario
  - London Regional Cancer Program, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario